CLINICAL TRIAL: NCT03621774
Title: Mobile-assisted Cognitive Behavioral Therapy for Negative Symptoms in Schizophrenia: An RCT
Brief Title: Mobile CBT for Negative Symptoms
Acronym: mCBTn
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Eric Granholm, Professor In Residence, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R33MH110019 (NIH)
Record Dates: First submitted 2018-08-03; First posted 2018-08-08 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-11

CONDITIONS: Schizophrenia; Schizoaffective Disorder
Keywords: Schizophrenia; CBT; Mobile CBT; Negative Symptoms
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mobile-assisted CBT-informed Skills Training (Experimental): Psychosocial intervention combining in-person and smartphone-based CBT-informed skills training for experiential negative symptoms in schizophrenia, called Mobile-assisted Cognitive-Behavioral Therapy for Negative symptoms (mCBTn).
  Interventions: Behavioral: Mobile-assisted CBT-informed Skills Training
- Supportive Contact (Placebo Comparator): An active group leader- and device-contact control group.
  Interventions: Behavioral: Supportive Contact

INTERVENTIONS:
Behavioral: Mobile-assisted CBT-informed Skills Training — mCBTn combines the CBT-informed components that target defeatist attitudes from Cognitive Behavioral Social Skills Training (CBSST) group skills training and mobile smartphone interventions from our prior clinical trials research.
  Arms: Mobile-assisted CBT-informed Skills Training
Behavioral: Supportive Contact — The SC intervention will provide the same amount of group and mobile device contact as the mCBTn condition. Participants will be carrying a phone but will not have access to the CBT-informed app. Group contact sessions will be semi-structured and consist of trouble-shooting device use and check-in about symptoms and potential crisis management, followed by a flexible discussion involving psychoeducation, instructions for accessing community crisis lines and related community resources, empathy, and non-directive reinforcement of health, coping, and symptom management behaviors that grow out of group discussions, with only minimal group leader guidance.
  Arms: Supportive Contact

SUMMARY:
This randomized controlled clinical trial will test a combined group contact plus mobile CBT-informed skills training intervention targeting defeatist attitudes in consumers with schizophrenia in comparison to a supportive contact control group in order to change motivational negative symptoms linked to defeatist attitudes.

DETAILED DESCRIPTION:
The primary purpose of this project is to determine if mCBTn at the optimal dose from the R61 produces greater reduction in severity of defeatist attitudes than a supportive contact control group in consumers with schizophrenia spectrum disorders with persistent moderate-to-severe experiential negative symptoms. A second aim is to determine whether reduction in defeatist attitudes mediates improvement in experiential negative symptoms and psychosocial functioning in mCBTn. The third aim is to determine whether mCBTn increases pupil dilation and whether changes in pupil dilation (an objective psychophysiological biomarker of effort) are associated with changes in defeatist attitudes and negative symptoms. The final aim is to explore predictors of response to mCBTn, including device use and group session adherence, demographics, neurocognitive impairment, and negative and other symptom severity at baseline.

ELIGIBILITY:
Inclusion Criteria:

* DSM-5 diagnosis of schizophrenia or schizoaffective disorder.
* Meets prospective criteria for persistent moderate-to-severe experiential negative symptoms in at least two of the three CAINS Motivation and Pleasure domains (mean of 2 -moderate- or greater for items averaged within the Social, Work or Recreational domains) at the beginning and end of a 2-week evaluation phase.
* Moderate-to-severe defeatist attitudes (DPAS > 50).
* ≥ 6th grade reading level on the Wide Range Achievement Test-4 Reading subtest (needed for reading treatment manual consumer workbook).
* Clinically stable and stable on current medications (no changes within 3 months prior to enrollment and meeting all inclusion/exclusion criteria during longitudinal baseline evaluation at both week -2 and 0).

Exclusion Criteria:

* Prior CBT in the past 2 years.
* Greater than moderate PANSS positive symptoms (P1-Delusions, P2- Disorganization, P3-Hallucinations, or P6-Suspiciousness - any item >5).
* Severe depression on the Calgary Depression Scale for Schizophrenia (CDS >8).
* Extrapyramidal symptoms.
* Ocular damage, disease, surgery or medications that affect pupil dilation.
* DSM-5 alcohol or substance use disorder in past 3 months.
* Level of care required interferes with outpatient skills training (e.g., hospitalized; severe medical illness).
* Unable to adequately see or manually manipulate the mobile device.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 112 (Actual)
Dates: Start 2019-03-27 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-08-31 (Actual)

PRIMARY OUTCOMES:
Defeatist performance beliefs (target mechanism) using the Defeatist Performance Attitude Scale | Assess change from baseline in defeatist performance beliefs at weeks 9, 18, and 42.
  Measure changes in defeatist performance beliefs severity using the Defeatist Performance Attitude Scale (DPAS). The DPAS is a 5-minute, 15-item self-report subscale derived from factor analysis of the commonly-used 40-item Dysfunctional Attitude Scale, which measures the tendency to overgeneralize from past failure experiences and form defeatist beliefs about the ability to perform future goal-directed tasks. Items are rated on a 1-7 Likert scale. A total score is reported with a range of 7 - 105 with higher total scores indicating more severe defeatist performance attitudes.
Clinical Assessment Interview for Negative Symptoms (CAINS) | Assess change from baseline in negative symptoms at weeks 9, 18, and 42.
  Measure changes in motivational negative symptoms on the CAINS. The CAINS is a 13-item interview-based assessment of negative symptoms, and each item is rated from 0 (no impairment) to 4 (severe deficit) measuring the two negative symptom factors recommended in consensus reports: Expression and Motivation and Pleasure (MAP) across social, vocational and recreational domains. Total scores for each factor are computed. The range for the MAP is 0 - 36, and the range for the Expression factor is 0 - 16. Higher scores indicate more severe negative symptoms for both factors.

SECONDARY OUTCOMES:
Pupillary responses as effort biomarker | Assess change from baseline in pupil dilation at weeks 9, 18, and 42.
  Measure changes in pupil dilation recorded during a digit span task.
Birchwood Social Functioning Scale (SFS) | Assess change from baseline in functioning at weeks 9, 18, and 42.
  Measure changes in functioning on the SFS. The SFS is a self-report assessment of functioning with 7 subscales, and each item is rated from 0 to 3 with the exception of the Occupation/Employment subscale if a participant is in regular employment (scores range from 7-10 based upon type of work). The subscales and score ranges are: Social Engagement Withdrawal (0-15), Interpersonal Communication/Relationships (0-30), Prosocial Activities (0-66), Recreation (0-48), Independence-Performance (0-39), Independence-Competence (0-39), and Occupation/Employment (0-10). Higher scores indicate better functioning for all subscales.

CONTACTS AND LOCATIONS:
Overall Officials: Eric Granholm, Ph.D., Principal Investigator — UC San Diego
Locations (1):
- UC San Diego, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Buchanan RW. Persistent negative symptoms in schizophrenia: an overview. Schizophr Bull. 2007 Jul;33(4):1013-22. doi: 10.1093/schbul/sbl057. Epub 2006 Nov 10. PMID 17099070
- [Background] Rector NA, Beck AT, Stolar N. The negative symptoms of schizophrenia: a cognitive perspective. Can J Psychiatry. 2005 Apr;50(5):247-57. doi: 10.1177/070674370505000503. PMID 15968839
- [Background] Granholm E, Ben-Zeev D, Link PC, Bradshaw KR, Holden JL. Mobile Assessment and Treatment for Schizophrenia (MATS): a pilot trial of an interactive text-messaging intervention for medication adherence, socialization, and auditory hallucinations. Schizophr Bull. 2012 May;38(3):414-25. doi: 10.1093/schbul/sbr155. Epub 2011 Nov 10. PMID 22080492
- [Background] Granholm E, Holden J, Link PC, McQuaid JR. Randomized clinical trial of cognitive behavioral social skills training for schizophrenia: improvement in functioning and experiential negative symptoms. J Consult Clin Psychol. 2014 Dec;82(6):1173-85. doi: 10.1037/a0037098. Epub 2014 Jun 9. PMID 24911420
- [Background] Granholm E, Ruiz I, Gallegos-Rodriguez Y, Holden J, Link PC. Pupillary Responses as a Biomarker of Diminished Effort Associated With Defeatist Attitudes and Negative Symptoms in Schizophrenia. Biol Psychiatry. 2016 Oct 15;80(8):581-8. doi: 10.1016/j.biopsych.2015.08.037. Epub 2015 Sep 15. PMID 26475673